CLINICAL TRIAL: NCT00492219
Title: Postoperative Function Following Partial and Total Knee Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer have access to equipment used for functional data collection
Sponsor: New Lexington Clinic (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Christian Christensen, MD, New Lexington Clinic, PSC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCO.2006.05
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2007-06

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis
Keywords: arthroplasty; replacement; knee; prosthesis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Patients undergoing total knee replacement
  Interventions: Device: Total Knee Replacement
- 2 (No Intervention): Healthy volunteers that are not undergoing knee replacement surgery
- 3 (Experimental): Patients undergoing partial knee replacement with the Oxford mobile bearing implant system
  Interventions: Device: Vanguard M fixed-bearing or Oxford mobile-bearing prostheses
- 4 (Experimental): Patients undergoing partial knee replacement with the Vanguard M implant system
  Interventions: Device: Vanguard M fixed-bearing or Oxford mobile-bearing prostheses

INTERVENTIONS:
Device: Vanguard M fixed-bearing or Oxford mobile-bearing prostheses — Patients that are appropriate for partial knee replacement will be randomized to receive one of these two FDA-approved implant systems.
  Other Names: All implant systems associated with this study are manufactured by Biomet, Inc. in Warsaw, IN.
  Arms: 3; 4
Device: Total Knee Replacement — Patients undergoing total knee replacement with the Vanguard Complete Knee implant system
  Other Names: All implant systems associated with this study are manufactured by Biomet, Inc. in Warsaw, IN.
  Arms: 1

SUMMARY:
The purpose of this study is to determine if patients with a fixed-bearing or mobile-bearing partial knee replacement perform functional activities differently than patients that have had total knee replacement or healthy volunteers that have not had knee surgery. The activities we are interested in include getting up out of a chair, stepping up and over a small wooden box, and standing still with the knees straight and also bent to 45 degrees.

DETAILED DESCRIPTION:
Patients will be asked for a brief medical history so that we may determine if he/she can participate in the study. If the patient is going to have partial knee replacement, he/she will be randomly assigned to receive either a fixed-bearing (Vanguard M, Biomet, Warsaw, IN) or mobile-bearing (Oxford, Biomet, Warsaw, IN) partial knee replacement. Both implant systems are FDA approved and Dr. Christensen is equally skilled with both systems. The fixed-bearing partial knee replacement is made up of a polished metal piece that is cemented to the femur and a metal piece that is cemented to the tibia. The plastic portion of the fixed-bearing partial knee replacement is attached to the tibial metal tray and does not move. The mobile-bearing knee replacement also has a metal pieces cemented to the femur and tibia, but between the two metal pieces is a small plastic piece that moves as the knee bends and straightens. Patients will have an equal opportunity of receiving either implant system.

If the patient is having total knee replacement, the surgery will be the same as if he/she did not participate in the study, except that we will collect information from the patient during office visits and will ask the patient to perform the functional tests. If the participant is one of the healthy volunteers, he/she will not have knee surgery and will only be asked to perform the functional tests.

Information collected during office visits:

A member of our research team will ask the patient a series of questions about the knee. Patients will be asked to answer this series of questions a total of 4 times over the course of 1 year. Also, we will record how well the patient can bend and straighten the knee at these 4 office visits. We will have patients rate the pain in their knee and ask if they are satisfied with the surgery. If patients have any complications, those will also be recorded. Patients will have X-rays taken of your knee at your follow-up visits. This is the normal routine following knee replacement. The X-rays will be read by the surgeon to help determine the success of the surgery.

We will also ask patients to perform 3 functional tests at each of these office visits. These 3 tests will be performed on a raised platform that is approximately 2 inches above the floor. For the first test, the patient will be asked to stand still with knees straight for two seconds, and then be asked to stand still with knees bent to 45 degrees for two seconds. For the second test, the patient will be asked to stand up from a seated position. For the third test, the patient will be asked to step up onto a four-inch wooden box and then step back down onto the platform. Prior to testing, the patient will be allowed to practice each of these tests as many times as necessary until he/she feels comfortable. During testing, an investigator will help make sure that the patient is able to safely and properly perform 3 repetitions of each test. We will not ask patients to perform one or more of the functional tests if they are unable to perform the test without constant use of their arms for support.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have elected to undergo either partial or total knee replacement, as well as a control group of patients free of lower extremity pathology

Exclusion Criteria:

* Sensory, neurological, or general health conditions that alter perception of the patient's limb in space
* Vestibular disorders will be excluded in order to protect against falls during functional testing
* Unable to understand the questions used to obtain the Knee Society Score
* Minors and prisoners will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Performance of three functional tests on a force platform | Baseline (preoperative), 6 weeks, 3 months, and 1, 2, and 5 years postoperative
Knee Society Scores | Baseline (preoperative), and 6 weeks, 3 months, and 1, 2, and 5 years after surgery
Patient Satisfaction | 6 weeks, 3 months, and 1, 2, and 5 years after surgery
Any postoperative complications | 6 weeks, 3 months, and 1, 2, and 5 years after surgery
Radiographic signs of component loosening or change of position, as well as progression of arthritis in the lateral compartment for the partial knee replacement patients | 6 weeks and 1, 2, and 5 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Christian P Christensen, MD, Principal Investigator — New Lexington Clinic
Locations (1):
- Lexington Clinic Sports Medicine Center, Lexington, Kentucky, United States

REFERENCES:
- [Background] Berend KR, Lombardi AV Jr. Liberal indications for minimally invasive oxford unicondylar arthroplasty provide rapid functional recovery and pain relief. Surg Technol Int. 2007;16:193-7. PMID 17429788
- [Background] Li MG, Yao F, Joss B, Ioppolo J, Nivbrant B, Wood D. Mobile vs. fixed bearing unicondylar knee arthroplasty: A randomized study on short term clinical outcomes and knee kinematics. Knee. 2006 Oct;13(5):365-70. doi: 10.1016/j.knee.2006.05.003. Epub 2006 Jun 22. PMID 16797994